CLINICAL TRIAL: NCT02272738
Title: A Phase I Study of Chemoradiotherapy Using Gemcitabine Plus Nab-paclitaxel for Unresectable Locally Advanced Pancreatic Adenocarcinoma
Brief Title: A Study of Chemoradiotherapy Using Gem Plus Nab-paclitaxel for Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Osaka Medical Center for Cancer and Cardiovascular Diseases (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TatsuyaIoka2013; UMIN 000012254 (Registry Identifier: UMIN)
Record Dates: First submitted 2014-10-18; First posted 2014-10-23 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Nab-Paclitaxel (Experimental): A conformal phase I study using 3 plus 3 method.
  Chemoradiotherapy while Gemcitabine, Nab-Paclitaxel are administered.
  Both Gemcitabine and Nab-Paclitaxel are an interventional agents in this arm.
  Gemcitabine is administered with 30 min intravenous infusion on day 1,8 and 15 every 4 weeks.
  Nab-Paclitaxel is administered with 30 min intravenous infusion on day 1,8 and 15 every 4 weeks.
  Radiotherapy (a total dose of 50.4Gy) was delivered in 28 fractions.
  Interventions: Drug: Gemcitabine; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine is administered with 30 min intravenous infusion on day 1,8 and 15 every 4 weeks.
  Other Names: Gemcitabine ；gemzer
Drug: Nab-Paclitaxel — Nab-Paclitaxel is administered with 30 min intravenous infusion on day 1,8 and 15 every 4 weeks.
  Other Names: Nab-Paclitaxel ；Abraxane

SUMMARY:
The purpose of this study is to evaluate the clinical safety and efficacy of Gemcitabine plus nab-Paclitaxel chemoradiotherapy and to determine the Maximal Tolerated Dose (MTD) for unresectable locally advanced pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Gemcitabine plus nab-Paclitaxel is one of the standard chemotherapy for metastatic pancreatic adenocarcinoma. Gemcitabine plus nab-Paclitaxel realize the favorable anti-tumor effect and tolerable toxicity. Gemcitabine plus nab-Paclitaxel is a promising regimen for concurrent chemoradiotherapy, but the investigators need to know the safety in the case of the concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced pancreatic cancer
* Locally advanced pancreatic cancer is defined as the presence of a surgically unresectable tumor(involving the celiac axis or the superior mesenteric artery)
* Performance Status:0-1(ECOG)
* Patients of age =>20 and 75>
* White Blood Cell (WBC) >=3,500/mm3,12,000/mm3,

  * Neutrophils >=1,500/mm3, platelets=100,000/mm3,
  * Hemoglobin >=9.5 g/dl,
  * GOT </=2.0 X Upper Limit Number (ULN),
  * Glutamate Pyruvate Transaminase (GPT) </=2.0 X ULN,
  * Alkaline Phosphatase (ALP) </=2.0 X ULN,
  * Total bilirubin <=1.5mg/dl,
  * Serum creatinine <=1.2mg/dl,
  * Creatinine clearance>=50 ml/min
  * arterial O2 pressure (PaO2) >=70torr or arterial O2 saturation (SpO2) >=96%
* Life expectancy more than 3 months.
* Written informed consent.

Exclusion Criteria:

* Active infection
* Lung fibrosis or intestinal pneumonia detectable on chest X-ray and CT
* Severe complication (heart disease, cirrhosis, diabetes)
* Myocardial infarction within 3 months
* Active synchronous or metachronous malignancy
* Pregnant or lactation women, or women with known or suspected pregnancy
* Symptomatic brain metastasis
* History of severe drug allergy
* Peripheral neuropathy
* Patients who are judged inappropriate for the entry into the study by the investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-08; Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with Adverse Events | 1 years

SECONDARY OUTCOMES:
Response Rate | 1 years
Overall Survival time | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuya Ioka, MD, Study Director — Osaka Medical Center for Cancer and Cardiovascular Diseases
Locations (1):
- Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Japan